CLINICAL TRIAL: NCT04919954
Title: Pharmacokinetics and Soft-Tissue Penetration of Tebipenem (SPR994) in Healthy Volunteer Subjects and Diabetic Patients With Lower Limb Infections
Brief Title: Tebipenem (SPR994) Tissue Penetration in Diabetic Patients With Wound Infections and Healthy Volunteers Via In Vivo Microdialysis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hartford Hospital (Other)
Collaborators: Spero Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: HHC-2021-0109
Record Dates: First submitted 2021-06-03; First posted 2021-06-09 (Actual); Last update posted 2023-10-23 (Actual); Status verified 2023-10

CONDITIONS: Diabetes; Wound Infection; ABSSSI; Healthy Volunteers
MeSH Terms: conditions — Diabetes Mellitus; Wound Infection

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Diabetic Wound Infection (Experimental): Participants with a documented medical history of Type 1 or Type 2 diabetes and a mild to moderate (Grade 2 or 3) wound infection of the lower limb will receive 3 to 7 doses of tebipenem, followed by sampling of interstitial tissue fluid at the margin of the wound by a microdialysis probe over 8 hours following the last dose.
  Interventions: Drug: Tebipenem Pivoxil Hydrobromide
- Healthy Volunteers (Active Comparator): Participants will be male or female healthy adult volunteers with no significant medical or medication history. Participants will receive 3 doses of tebipenem, followed by sampling of interstitial tissue fluid by a microdialysis probe inserted in a thigh over 8 hours following the last dose.
  Interventions: Drug: Tebipenem Pivoxil Hydrobromide

INTERVENTIONS:
Drug: Tebipenem Pivoxil Hydrobromide — Tebipenem 300 mg or 600 mg will be administered orally every 8 hours for total of 3 to 7 doses

SUMMARY:
This study will determine the tissue penetration of a broad-spectrum orally bioavailable carbapenem, tebipenem pivoxil hydrobromide (SPR994) (Spero Therapeutics, Inc.), into the extracellular, interstitial fluid of soft tissue in diabetic patients with lower limb wound infections. Penetration will be compared with a group of healthy volunteer control participants.

DETAILED DESCRIPTION:
This study will enroll 10 patients with diabetes who are admitted with a lower limb wound infection and 6 healthy volunteer control participants. The study will take place in an inpatient unit at Hartford Hospital for all patients and in the Clinical Research Center at Hartford Hospital for all healthy volunteers. All participants will receive 3 to 7 doses of tebipenem pivoxil hydrobromide (300 mg or 600 mg orally every 8 hours depending on renal function). A microdialysis probe (Mdialysis Inc., N. Chelmsford, MA) will be inserted into the subcutaneous soft tissue near the margin of the wound (patients) or in the thigh (healthy volunteers). The microdialysis probe is perfused with normal saline solution and samples are collected for the 8 hours following the final dose. A peripheral intravenous catheter will be inserted into an arm vein to collect blood samples simultaneously with microdialysis samples. Concentrations in tissue are compared with blood to determine percent penetration.

ELIGIBILITY:
Exclusion Criteria - All patients/participants

Participants in the diabetic wound group or healthy volunteer group will be excluded if any of the following criteria are met:

1. Less than 18 years of age
2. History of hypersensitivity or allergy to tebipenem or its derivatives and any β-lactam antibiotic
3. History of hypersensitivity to lidocaine or lidocaine derivatives
4. Concurrently receiving probenecid.
5. Males who are not surgically sterilized (with female partners of childbearing potential) and females of childbearing potential must agree to use two highly effective methods of contraception from screening, during this trial, and for 90 days after the last dose of study drug. A woman is considered of childbearing potential unless postmenopausal (≥1 year without menses) or surgically sterilized via bilateral oophorectomy, hysterectomy, bilateral tubal ligation, or successful Essure® placement with a documented confirmation test at least 90 days after the procedure. Highly effective contraception is defined as a method of contraception that has a less than 1% failure rate when used consistently and correctly. These methods are as follows:

   * Hormonal contraceptives (eg, combined oral contraceptives, patch, vaginal ring, injectables, and implants).
   * Intrauterine device or intrauterine system.
   * Double-barrier methods of contraception (eg, male condom with diaphragm or male condom with cervical cap).
   * Monogamous relationship with a vasectomized partner.
   * Total abstinence, in accordance with the lifestyle of the subject.
6. Any other documented reason felt by the investigator to potentially affect the outcomes of the study

Additional Exclusion Criteria for Diabetic Patient Study Group

1. Participants likely to require multiple surgical interventions during the study period, which could affect placement of the microdialysis catheter
2. Creatinine clearance (CrCl) < 30ml/min, as calculated by Cockroft-Gault using ideal body weight

Additional Exclusion Criteria for Healthy Volunteer Control Group

1. Body Mass Index (BMI) ≥ 35 kg/m2
2. Creatinine clearance (CrCl) < 50ml/min, as calculated by Cockroft-Gault using ideal body weight
3. Presence of anemia, thrombocytopenia, or leukopenia as defined by hematocrit, platelet, or white blood cell count < 75% of the lower limit of normal
4. Aspartate transaminase, alanine aminotransferase, or alkaline phosphatase greater than five times upper limit of normal
5. Total bilirubin greater than three times the upper limit of normal
6. Any known active co-morbidity listed on medical history or that becomes apparent during physical examination
7. Positive urine drug screen (cocaine, THC, opiates, benzodiazepines, and amphetamines)
8. History of regular alcohol consumption exceeding 7 drinks/week for females or 14 drinks/week for men (1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor) within 6 months of screening.
9. Use of tobacco- or nicotine-containing products in excess of the equivalence of 5 cigarettes per day.
10. Consumption of caffeine between Study Days -1 and 2.
11. Use of prescription or non-prescription drugs, vitamins, or dietary supplements within 7 days or 5 half-lives (whichever is longer) prior to the first dose of study medication, with the exception of acetaminophen at doses of ≤ 1 g/day. The use of hormonal methods of contraception (including oral and transdermal contraceptives, injectable progesterone, progestin subdermal implants, progesterone-releasing IUDs, postcoital contraceptive methods) are permitted.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-07-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-12-23 (Actual)

PRIMARY OUTCOMES:
Tebipenem Pivoxil Hydrobromide Tissue Penetration | 8 hours
  The ratio of tebipenem tissue concentrations to blood concentrations following the final tebipenem dose

SECONDARY OUTCOMES:
Tebipenem Pivoxil Hydrobromide Area Under the Curve (AUC) in Tissue | 8 hours
  The area under the drug concentration-time curve (AUC) in tissue reflects the actual tissue exposure to drug after administration of a dose of the drug and is expressed in mg*h/L. Venous blood will be obtained via peripheral intravenous catheter immediately before administration of the last dose (pre-dose timepoint), and at 9 time-points post-dose. Dialysate samples of 120μL will be collected in 200µL microvials simultaneously with plasma samples.

CONTACTS AND LOCATIONS:
Overall Officials: Tomefa E Asempa, PharmD, Principal Investigator — Hartford Hospital
Locations (1):
- Hartford Hospital, Hartford, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No